CLINICAL TRIAL: NCT07059429
Title: Randomized Controlled Study of Ketamine Administration for Postoperative Pain Management in Patients Undergoing Knee Arthroplasty,
Brief Title: Ketamine Administration for Postoperative Pain Management in Patients Undergoing Knee Arthroplasty
Acronym: KETARTHRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMSC-01-25
Record Dates: First submitted 2025-07-07; First posted 2025-07-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Knee Arthroplasty; Postoperative Pain; Pain Management; Analgesia; Opioid Use; Ketamine
Keywords: Ketamine; Knee Replacement; Total Knee Arthroplasty; Postoperative Analgesia; Patient-Controlled Analgesia; PCA; Opioid Sparing; Multimodal Pain Management; Morphine Consumption; Neuropsychiatric Side Effects; Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Nausea; Vomiting | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups:
  the intervention group (standardized postoperative analgesia plus ketamine infusion via patient-controlled analgesia),
  or the control group (standardized postoperative analgesia without ketamine). Randomization will be performed using permuted blocks of six patients. There will be no crossover or switching between groups; all interventions and assessments will be conducted independently and concurrently for both groups.
  The study is single-center and prospective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine Plus Standard Analgesia (Experimental): Participants in this group will receive standardized postoperative pain management (ketoprofen 100 mg twice daily and paracetamol 1000 mg every 8 hours for 24 hours after knee arthroplasty) plus a continuous intravenous infusion of ketamine using PCA at 0.15 mg/kg/h, with 1 mg boluses available every 5 minutes (maximum daily dose 500 mg), for 24 hours after knee arthroplasty. Morphine 10 mg intramuscularly (IM) may be administered as needed for rescue therapy.
  Interventions: Drug: Ketamine
- Standard Analgesia Alone (Active Comparator): Participants in this group will receive standardized postoperative pain management (ketoprofen 100 mg twice daily and paracetamol 1000 mg every 8 hours for 24 hours after knee arthroplasty) without ketamine infusion. Morphine 10 mg IM may be administered as needed for rescue therapy.
  Interventions: Drug: Standard Analgesia

INTERVENTIONS:
Drug: Ketamine — Ketamine administered intravenously at 0.15 mg/kg/h via PCA with 1 mg boluses, 5-minute lockout, maximum 500 mg per 24 hours after knee arthroplasty.
  Arms: Ketamine Plus Standard Analgesia
Drug: Standard Analgesia — Standard analgesia includes ketoprofen 100 mg twice daily and paracetamol 1000 mg every 8 hours for 24 hours after knee arthroplasty; morphine 10 mg IM as needed for rescue therapy.
  Arms: Standard Analgesia Alone

SUMMARY:
This study is conducted to evaluate the effectiveness and safety of ketamine infusion for pain relief after knee replacement surgery. Adult patients who have undergone knee arthroplasty will be randomly assigned to one of two groups. The study group will receive standard pain management plus a continuous infusion of ketamine using patient-controlled analgesia (PCA), while the control group will only receive standard pain management. All patients will be monitored for pain intensity using the Numeric Rating Scale (NRS) at several time points the first 24 hours after surgery. The study will compare the total amount of opioid pain medication required, the level of pain experienced, and the frequency and severity of side effects such as nausea, vomiting, and neuropsychiatric reactions. The goal is to determine whether adding ketamine to standard pain management reduces opioid use and improves pain control without increasing side effects. The results improve pain management strategies after knee replacement surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled study evaluating the use of ketamine infusion as part of postoperative pain management for adult patients undergoing knee arthroplasty. The study will enroll patients aged 18 to 90 years who have undergone knee replacement surgery at the N.I. Pirogov National Medical and Surgical Center.

Participants will be randomly assigned to either the study group or the control group. Both groups will receive standardized pain management with ketoprofen and paracetamol in keeping with current guidelines. The study group will receive an additional continuous infusion of ketamine using PCA at a rate of 0.15 mg/kg/h, with 1 mg boluses available in 5-minute lockout intervals and a maximum daily dose of 500 mg. In both groups, opioid analgesics (morphine 10 mg intramuscularly as needed) will be administered if pain control is inadequate. Regional nerve blocks may be repeated under ultrasound guidance if necessary; patients requiring repeated femoral nerve block will be analyzed separately.

Pain intensity will be assessed using the NRS at 0, 2, 4, 6, 10, 14, 18, and 24 hours postoperatively. Data will be collected on the total dose of opioids used, additional analgesic requirements, the number and severity of neuropsychiatric adverse events (graded according to CTCAE), the frequency of postoperative nausea and vomiting, and the total dose and number of ketamine boluses administered.

The primary outcome is the total dose of opioid analgesics (morphine equivalents, mg) administered the first 24 hours after surgery. Secondary outcomes include pain scores at each time point, incidence and severity of neuropsychiatric side effects, frequency of postoperative nausea and vomiting, and total ketamine dose received.

The study is designed to compare the efficacy and safety of ketamine infusion in reducing opioid consumption and improving pain control after knee arthroplasty, while closely monitoring adverse events. The results aim to provide evidence for optimizing multimodal analgesia in orthopedic surgery.This clinical trial was preceded by a pilot study involving patients undergoing knee arthroplasty. The pilot phase aimed to evaluate the variability of key parameters such as pain intensity, opioid requirements, and the incidence of neuropsychiatric side effects. Based on the analysis of the investigators' published data, modifications were made in the main study protocol, including adjustments to the ketamine bolus dose within the PCA regimen to optimize efficacy and safety.

The changes were introduced to enhance pain control and minimize adverse effects in the main study population. The current trial involves these protocol refinements, and the investigators anticipate that the optimized ketamine dosing schedule will lead to improved outcomes compared to the initial regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years and less than 90 years.
* Patients who have undergone knee arthroplasty.
* The patient has read the information sheet and signed the informed consent form.

Exclusion Criteria:

* Spinal anesthesia performed intraoperatively.
* Epidural analgesia administered postoperatively.
* Perioperative blockade of the sciatic nerve, genicular nerve, or lumbar plexus.
* Allergy to ketamine or non-steroidal anti-inflammatory drugs.
* Contraindications to ketamine as specified in the product instructions.
* Time from the end of surgery to study enrollment exceeds 24 hours.
* Ineffectiveness of analgesia as provided by the study protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Consumption in Morphine Equivalents Within 24 Hours After Surgery | 24 hours postoperatively
  The total dose of opioid analgesics (calculated in milligrams of morphine equivalents) administered to each patient during the first 24 hours after knee arthroplasty.

SECONDARY OUTCOMES:
Pain Intensity Assessed by Numeric Rating Scale (NRS) | At 0, 2, 4, 6, 10, 14, 18, and 24 hours postoperatively
  Pain intensity scores measured using the NRS at specified time points (0, 2, 4, 6, 10, 14, 18, 24 hours after surgery). The NRS is an 11-point scale ranging from 0 to 10, where:
  0 corresponds to "no pain," 10 corresponds to "the worst pain imaginable."
Incidence of Postoperative Nausea and Vomiting | 24 hours postoperatively
  The number of patients experiencing any episode of postoperative nausea or vomiting during the first 24 hours after surgery.
Incidence of Neuropsychiatric Adverse Events | 24 hours postoperatively
  The number of patients experiencing one or more neuropsychiatric adverse events (such as hallucinations, agitation, or dysphoria) during the first 24 hours postoperatively.
Severity of Neuropsychiatric Adverse Events | 24 hours postoperatively
  The maximum severity of any neuropsychiatric adverse event experienced by a patient, graded according to the Common Terminology Criteria for Adverse Events (CTCAE). The scale ranges from Grade 1 (Mild) to Grade 5 (Death). Specific conditions and symptoms may have values or descriptive comment for each level, but the general guideline is:
  1. - Mild
  2. - Moderate
  3. - Severe
  4. - Life-threatening
  5. - Death
Total Number of Ketamine Boluses Administered | 24 hours postoperatively
  The total count of patient-initiated ketamine boluses administered via Patient-Controlled Analgesia (PCA) during the first 24 hours after surgery.
Cumulative Ketamine Dose Administered | 24 hours postoperatively
  The total cumulative dose of ketamine (in milligrams) administered during the first 24 hours after surgery, including both the continuous infusion and patient-initiated boluses.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Teplykh, MD, Study Director — Pirogov National Medical and Surgical Center; Ivan Shcheparev, MD, PhD, Principal Investigator — Pirogov National Medical and Surgical Center
Locations (1):
- Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 2 months after completion of the study
Access Criteria: upon the request

REFERENCES:
- [Background] Laskowski K, Stirling A, McKay WP, Lim HJ. A systematic review of intravenous ketamine for postoperative analgesia. Can J Anaesth. 2011 Oct;58(10):911-23. doi: 10.1007/s12630-011-9560-0. Epub 2011 Jul 20. PMID 21773855
- [Background] Subramaniam K, Subramaniam B, Steinbrook RA. Ketamine as adjuvant analgesic to opioids: a quantitative and qualitative systematic review. Anesth Analg. 2004 Aug;99(2):482-95, table of contents. doi: 10.1213/01.ANE.0000118109.12855.07. PMID 15271729
- [Background] Guillou N, Tanguy M, Seguin P, Branger B, Campion JP, Malledant Y. The effects of small-dose ketamine on morphine consumption in surgical intensive care unit patients after major abdominal surgery. Anesth Analg. 2003 Sep;97(3):843-847. doi: 10.1213/01.ANE.0000075837.67275.36. PMID 12933413
- [Background] Jouguelet-Lacoste J, La Colla L, Schilling D, Chelly JE. The use of intravenous infusion or single dose of low-dose ketamine for postoperative analgesia: a review of the current literature. Pain Med. 2015 Feb;16(2):383-403. doi: 10.1111/pme.12619. Epub 2014 Dec 19. PMID 25530168
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Fischer HB, Simanski CJ, Sharp C, Bonnet F, Camu F, Neugebauer EA, Rawal N, Joshi GP, Schug SA, Kehlet H; PROSPECT Working Group. A procedure-specific systematic review and consensus recommendations for postoperative analgesia following total knee arthroplasty. Anaesthesia. 2008 Oct;63(10):1105-23. doi: 10.1111/j.1365-2044.2008.05565.x. Epub 2008 Jul 10. PMID 18627367
- [Background] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Background] Bell RF, Dahl JB, Moore RA, Kalso EA. WITHDRAWN: Perioperative ketamine for acute postoperative pain. Cochrane Database Syst Rev. 2015 Jul 2;2015(7):CD004603. doi: 10.1002/14651858.CD004603.pub3. PMID 26133677
- [Background] Porter SB, McClain RL, Howe BL, Ardon AE, Mazer LS, Knestrick BM, Clendenen AM. Perioperative ketamine for acute postoperative analgesia: the Mayo Clinic-Florida experience. J Perianesth Nurs. 2015 Jun;30(3):189-95. doi: 10.1016/j.jopan.2015.01.010. PMID 26003764
- [Background] Pouldar TM, Maher DP, Betz AW, Wiegers JJ, Friedman JA, Zaidi SS, Rejali A, Tran HP, Yumul R, Louy C. Adverse Effects Associated with Patient-Controlled Analgesia with Ketamine Combined with Opioids and Ketamine Infusion with PCA Bolus in Postoperative Spine Patients: A Retrospective Review. J Pain Res. 2022 Oct 10;15:3127-3135. doi: 10.2147/JPR.S358770. eCollection 2022. PMID 36247824
- [Background] Seman MT, Malan SH, Buras MR, Butterfield RJ, Harold KL, Madura JA, Rosenfeld DM, Gorlin AW. Low-Dose Ketamine Infusion for Perioperative Pain Management in Patients Undergoing Laparoscopic Gastric Bypass: A Prospective Randomized Controlled Trial. Anesthesiol Res Pract. 2021 Jul 21;2021:5520517. doi: 10.1155/2021/5520517. eCollection 2021. PMID 34335740
- [Background] Puzio TJ, Klugh J, Wandling MW, Green C, Balogh J, Prater SJ, Stephens CT, Sergot PB, Wade CE, Kao LS, Harvin JA. Ketamine for acute pain after trauma: the KAPT randomized controlled trial. Trials. 2022 Jul 27;23(1):599. doi: 10.1186/s13063-022-06511-6. PMID 35897081
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- See also: Official website of the Pirogov National Medical and Surgical Center — https://www.pirogov-center.ru/english/about/